CLINICAL TRIAL: NCT00092547
Title: A Safety and Immunogenicity Study of Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in Preadolescents and Adolescents (Base Study). A Long Term Immunogenicity, Safety, and Effectiveness Study of GARDASIL (Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine) Among Adolescents Who Received GARDASIL at 9-18 Years of Age (Extension Study).
Brief Title: A Study of Gardasil (V501) in Preadolescents and Adolescents (V501-018)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-018; 2004_084
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Results first posted 2010-05-04 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Human; Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- qHPV Vaccine in Base Study (Experimental): Represents participants who were randomized into the qHPV Group, who received three 0.5 mL intramuscular injections of V501 (qHPV) at Day 1, Month 2, and Month 6.
  Interventions: Biological: V501
- Placebo in Base Study (Placebo Comparator): Represents participants who were randomized into the Placebo Group, who received three 0.5 mL intramuscular injections of placebo at Day 1, Month 2, and Month 6.
  Interventions: Biological: Comparator: Placebo
- qHPV Vaccine in Extension Study (Experimental): Represents participants originally enrolled into the Placebo Group who continued in the study to receive 0.5 mL intramuscular injections of V501 (qHPV) at Month 30, Month 32, and Month 36.
  Interventions: Biological: V501

INTERVENTIONS:
Biological: V501 — 0.5 mL intramuscular injection of V501
  Other Names: GARDASIL™
  Arms: qHPV Vaccine in Base Study; qHPV Vaccine in Extension Study
Biological: Comparator: Placebo — 0.5 mL intramuscular injection of placebo
  Arms: Placebo in Base Study

SUMMARY:
This study is to evaluate the safety, tolerability, and immune response of an investigational vaccine in preadolescent and adolescent boys and girls for the prevention of Human Papilloma Virus (HPV).

DETAILED DESCRIPTION:
The original base protocol (V501-018)(NCT00092547) was extended in amendments V501-018-05 and -06 to provide 37 months of follow-up. Additionally, subjects in the Placebo Group during the base study were given 3 doses of open-label GARDASIL™ (V501) at Months 30, 32, and 36.

The study was extended again in amendment V501-018-10(NCT00092547), titled "A Long Term Immunogenicity, Safety, and Effectiveness Study of GARDASIL (Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine) Among Adolescents Who Received GARDASIL at 9-18 Years of Age" to allow a follow-up period to Month 126.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents and preadolescents with no prior sexual history

Exclusion Criteria:

* Subjects with compromised immune system or have a history of severe allergic reaction

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1781 (Actual)
Dates: Start 2003-10-08 (Actual); Primary Completion 2005-11-03 (Actual); Study Completion 2015-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Reisinger KS, Block SL, Lazcano-Ponce E, Samakoses R, Esser MT, Erick J, Puchalski D, Giacoletti KE, Sings HL, Lukac S, Alvarez FB, Barr E. Safety and persistent immunogenicity of a quadrivalent human papillomavirus types 6, 11, 16, 18 L1 virus-like particle vaccine in preadolescents and adolescents: a randomized controlled trial. Pediatr Infect Dis J. 2007 Mar;26(3):201-9. doi: 10.1097/01.inf.0000253970.29190.5a. PMID 17484215
- [Background] Perez G, Lazcano-Ponce E, Hernandez-Avila M, Garcia PJ, Munoz N, Villa LL, Bryan J, Taddeo FJ, Lu S, Esser MT, Vuocolo S, Sattler C, Barr E. Safety, immunogenicity, and efficacy of quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like-particle vaccine in Latin American women. Int J Cancer. 2008 Mar 15;122(6):1311-8. doi: 10.1002/ijc.23260. PMID 18000825
- [Result] Ferris D, Samakoses R, Block SL, Lazcano-Ponce E, Restrepo JA, Reisinger KS, Mehlsen J, Chatterjee A, Iversen OE, Sings HL, Shou Q, Sausser TA, Saah A. Long-term study of a quadrivalent human papillomavirus vaccine. Pediatrics. 2014 Sep;134(3):e657-65. doi: 10.1542/peds.2013-4144. Epub 2014 Aug 18. PMID 25136050
- [Result] Ferris DG, Samakoses R, Block SL, Lazcano-Ponce E, Restrepo JA, Mehlsen J, Chatterjee A, Iversen OE, Joshi A, Chu JL, Krick AL, Saah A, Das R. 4-Valent Human Papillomavirus (4vHPV) Vaccine in Preadolescents and Adolescents After 10 Years. Pediatrics. 2017 Dec;140(6):e20163947. doi: 10.1542/peds.2016-3947. PMID 29167376
- [Derived] Garland SM, Ault KA, Gall SA, Paavonen J, Sings HL, Ciprero KL, Saah A, Marino D, Ryan D, Radley D, Zhou H, Haupt RM, Garner EIO; Quadrivalent Human Papillomavirus Vaccine Phase III Investigators. Pregnancy and infant outcomes in the clinical trials of a human papillomavirus type 6/11/16/18 vaccine: a combined analysis of five randomized controlled trials. Obstet Gynecol. 2009 Dec;114(6):1179-1188. doi: 10.1097/AOG.0b013e3181c2ca21. PMID 19935017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1781 participants were randomized to receive qHPV or Placebo in the Base Study. At month 30, participants who received Placebo in the Base Study were eligible to receive qHPV, and formed the Extension Group. Participants were to be followed for safety and efficacy for up to 10 years.
Groups:
- qHPV Vaccine in Extension Study: Represent participants originally enrolled into the Placebo Group who continued in the study to receive 0.5 mL intramuscular injections of V501 (qHPV) at Month 30, Month 32, and Month 36.
Period: Base Vaccine Phase (Day 1 to Month 7)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 1184 | 597 | 0
Vaccinated | 1179 | 596 | 0
Completed | 1121 | 561 | 0
Not Completed | 63 | 36 | 0
Not completed — Not Vaccinated | 5 | 1 | 0
Not completed — Adverse Event | 4 | 1 | 0
Not completed — Lost to Follow-up | 18 | 7 | 0
Not completed — Withdrawal by Subject | 28 | 21 | 0
Not completed — Moved | 3 | 1 | 0
Not completed — per sponsor request: (noncompliant) | 0 | 1 | 0
Not completed — Did not meet local regulations | 0 | 1 | 0
Not completed — Refused Vaccination | 5 | 3 | 0
Period: Base Follow-up Phase (Month 7 to 18)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 1128 (Includes participants continuing and who previously discontinued who re-entered the study) | 565 (Includes participants continuing and who previously discontinued who re-entered the study) | 0
Completed | 1108 | 551 | 0
Not Completed | 20 | 14 | 0
Not completed — Subject moved | 1 | 5 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0
Not completed — Lost to Follow-up | 13 | 7 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Base Follow-up Phase (Month 18 to 30)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 964 (Includes participants continuing and who previously discontinued who re-entered the study) | 490 (Includes participants continuing and who previously discontinued who re-entered the study) | 0
Completed | 956 | 485 | 0
Not Completed | 8 | 5 | 0
Not completed — Subject moved | 4 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Extension Vaccine Phase (Month 30 to 37)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 956 (Includes participants continuing and who previously discontinued who re-entered the study) | 0 | 485 (Includes participants continuing and who previously discontinued who re-entered the study)
Vaccinated in Extension Study | 0 | 0 | 482
Completed | 933 | 0 | 469
Not Completed | 23 | 0 | 16
Not completed — Subject moved | 3 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 9
Not completed — Lost to Follow-up | 14 | 0 | 7
Period: Long-term Follow-up (Month 42 Visit)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 612 (Includes participants continuing and who previously discontinued who re-entered the study) | 0 | 308 (Includes participants continuing and who previously discontinued who re-entered the study)
Completed | 611 | 0 | 308
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Long-term Follow-up (Month 72 Visit)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 550 (Includes participants continuing and who previously discontinued who re-entered the study) | 0 | 276 (Includes participants continuing and who previously discontinued who re-entered the study)
Completed | 550 | 0 | 276
Not Completed | 0 | 0 | 0
Period: Long-term Follow-up (Month 96 Visit)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 508 (Includes participants continuing and who previously discontinued who re-entered the study) | 0 | 267 (Includes participants continuing and who previously discontinued who re-entered the study)
Completed | 508 | 0 | 267
Not Completed | 0 | 0 | 0
Period: Long-term Follow-up (Month 126 Visit)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | qHPV Vaccine in Extension Study
Started | 454 | 0 | 211
Completed | 454 | 0 | 211
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | Total
Number analyzed (Participants) | 1184 | 597 | 1781
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (1.9) | 11.8 (1.9) | 11.9 (1.9)
Age, Customized [Number; unit: Participants]
  8 Years of Age and Under | 0 | 0 | 0
  9 to 16 Years of Age | 1184 | 597 | 1781
  17 Years of Age and Over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 616 | 322 | 938
  Male | 568 | 275 | 843
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 149 | 70 | 219
  Black | 50 | 21 | 71
  Hispanic American | 260 | 130 | 390
  Native American | 0 | 1 | 1
  White | 716 | 369 | 1085
  Other | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Experiences (SAEs) Through Month 18
Description: Tolerability as assessed by the number of participants with clinical adverse experiences through Month 18. A serious adverse event is any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgment.
Time Frame: Up to Month 18
Population: All participants who were vaccinated according to actual treatment received (qHPV or placebo) and had safety follow-up.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1165 | 584
participants | 6 | 0

2. Primary Outcome: Number of Participants Reporting SAEs From Month 18 Through Month 37
Description: Tolerability as assessed by the number of participants with clinical adverse experiences from Month 18 through Month 37
Time Frame: Month 18 to Month 37
Population: All participants who were vaccinated according to actual treatment received (qHPV or placebo) and had safety follow-up.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 923 | 477
participants | 0 | 3

3. Primary Outcome: Number of Participants Reporting Other (Non-serious) AEs Through Month 18
Description: Tolerability as assessed by the number of participants with clinical adverse experiences through Month 18
Time Frame: Up to Month 18: Injection site AEs were collected from Days 1-5 and other non-serious AEs from Days 1-15 after any vaccination
Population: All participants who were vaccinated according to actual treatment received (qHPV or placebo) and had safety follow-up.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1165 | 584
participants | 918 | 340

4. Primary Outcome: Percentage of Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 72
Description: A participant is considered seropositive for a given HPV type if he or she has a cLIA titer at or above the serostatus cutoff for that HPV type. Serostatus cutoffs are ≥ 20 mMU/mL for HPV 6 and 16, ≥ 16 mMU/mL for HPV 11, and ≥ 24 mMU/mL for HPV 18.
Time Frame: Month 72 (66 Months Post-dose 3 for the Original qHPV Vaccine Cohort and 36 months Post-dose 3 for the Extension Group)
Population: Per-protocol population: participants without protocol violations who received all 3 vaccinations, were seronegative to the respective HPV type at Day 1 (for the Base Vaccination group), or Month 30 (for the Extension Group), and had a valid serology result at the specified time for assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 550 | 276
Percentage of participants
  Type 6: n=475, 151 | 93.3 [90.6 to 95.3] | 91.4 [85.7 to 95.3]
  Type 11: n=475, 151 | 96.0 [93.8 to 97.6] | 96.7 [92.4 to 98.9]
  Type 16: n=473, 154 | 97.9 [96.1 to 99.0] | 97.4 [93.5 to 99.3]
  Type 18: n=477, 160 | 74.4 [70.3 to 78.3] | 79.4 [72.3 to 85.4]

5. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 6, 11, 16, and 18 at Month 72
Time Frame: Month 72 (66 Months Post-dose 3 for the Original qHPV Vaccine Cohort and 36 months Post-dose 3 for the Extension Group)
Population: Per-protocol population: participants without protocol violations who received all 3 vaccinations within appropriate day ranges as defined in the CSR, were seronegative to the respective HPV type at Day 1 (for the Main Vaccination group), or Month 30 (for the Extension Group), and had a valid serology result at the specified time for assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 550 | 276
milliMerck units/mL
  Type 6: n=475, 151 | 118.9 [108.4 to 130.4] | 113.9 [95.7 to 135.6]
  Type 11: n=475, 151 | 135.7 [122.6 to 150.3] | 137.9 [114.9 to 165.5]
  Type 16: n=473, 154 | 521.2 [466.2 to 582.6] | 485.8 [396.4 to 595.3]
  Type 18: n=477, 160 | 70.9 [61.8 to 81.4] | 67.7 [53.1 to 86.3]

6. Primary Outcome: Geometric Mean Titers for Anti-HPV 6, 11, 16, and 18 at Month 96
Time Frame: Month 96 (90 Months Post-dose 3 for Original qHPV Vaccine Group and 60 Months Post-dose 3 for Extension Group)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 508 | 267
milliMerck units/mL
  Type 6: n=451, 141 | 71.4 [64.6 to 79.0] | 91.0 [76.4 to 108.6]
  Type 11: n=451, 141 | 67.5 [60.1 to 75.7] | 90.3 [74.0 to 110.1]
  Type 16: n=447, 143 | 325.5 [288.6 to 367.1] | 387.4 [314.7 to 476.9]
  Type 18: n=452, 152 | 41.6 [36.5 to 47.5] | 48.3 [37.6 to 62.0]

7. Primary Outcome: Percentage of Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 96
Description: as for outcome 4
Time Frame: Month 96 (90 Months Post-dose 3 for Original qHPV Vaccine Cohort and 60 Months Post-dose 3 for Extension Group)
Population: Per-protocol population: participants without protocol violations who received all 3 qHPV vaccinations, were seronegative to the respective HPV type at Day 1 (for the Main Vaccination group), or Month 30 (for the Extension Group), and had a valid serology result at the specified time for assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 508 | 267
Percentage of participants
  Type 6: n=451, 141 | 88.2 [84.9 to 91.1] | 91.5 [85.6 to 95.5]
  Type 11: n=451, 141 | 89.1 [85.9 to 91.9] | 93.6 [88.2 to 97.0]
  Type 16: n=447, 143 | 96.9 [94.8 to 98.3] | 97.9 [94.0 to 99.6]
  Type 18: n=452, 152 | 63.9 [59.3 to 68.4] | 69.1 [61.1 to 76.3]

8. Primary Outcome: Geometric Mean Titers for Anti-HPV 6, 11, 16, and 18 at Month 126
Time Frame: Month 126 (120 Months Post-dose 3 for Original qHPV Vaccine Cohort and 90 Months Post-dose 3 for Extension Group)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 454 | 211
milliMerck units/mL
  Type 6: n=409, 112 | 88.0 [78.9 to 98.2] | 99.3 [81.0 to 121.6]
  Type 11: n=409, 112 | 74.6 [66.1 to 84.1] | 96.0 [76.1 to 121.1]
  Type 16: n=403, 115 | 320.1 [281.2 to 364.4] | 351.6 [277.1 to 446.2]
  Type 18: n=408, 120 | 36.5 [31.7 to 42.1] | 39.6 [30.7 to 51.2]

9. Primary Outcome: Percentage of Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 126
Description: as for outcome 4
Time Frame: Month 126 (120 Months Post-dose 3 for Original qHPV Vaccine Cohort and 90 Months Post-dose 3 for Extension Group)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 454 | 211
Percentage of participants
  Type 6: n=409, 112 | 89.0 [85.6 to 91.9] | 91.1 [84.2 to 95.6]
  Type 11: n=409, 112 | 88.8 [85.3 to 91.6] | 92.9 [86.4 to 96.9]
  Type 16: n=403, 115 | 96.0 [93.6 to 97.7] | 96.5 [91.3 to 99.0]
  Type 18: n=408, 120 | 60.5 [55.6 to 65.3] | 65.0 [55.8 to 73.5]

10. Primary Outcome: Number of Participants Reporting SAEs Related to Study Vaccine or to a Study Procedure in the Long-term Follow-up
Description: A serious adverse event is any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgment. SAEs considered by the investigator to be possibly, probably, or definitely related to study vaccine or a study procedure were reported.
Time Frame: Month 37 to Month 126
Population: The analysis population was all participants who were vaccinated according to actual treatment received and had safety follow-up.
Measure: Number; unit: Participants
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 821 | 424
Participants | 0 | 1

11. Secondary Outcome: Percentage of Original qHPV Vaccine Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 1 Postdose 3 (Month 7)
Description: as for outcome 4
Time Frame: Month 7 (1 Month Postdose 3)
Population: Per-protocol population: participants without protocol violations who received all 3 qHPV vaccinations, were seronegative to the respective HPV type at Day 1, and had a valid serology result at the specified time for assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 1082
Percentage of participants
  Type 6: n=953 | 99.8 [99.2 to 100]
  Type 11: n=954 | 99.8 [99.2 to 100]
  Type 16: n=949 | 99.7 [99.1 to 99.9]
  Type 18: n=956 | 99.7 [99.1 to 99.9]

12. Secondary Outcome: Percentage of Original qHPV Vaccine Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 12 Postdose 3 (Month 18).
Description: as for outcome 4
Time Frame: Month 18 (12 Months Post-dose 3)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 1106
Percentage of participants
  Type 6: n=937 | 97.8 [96.6 to 98.6]
  Type 11: n=938 | 99.3 [98.5 to 99.7]
  Type 16: n=933 | 99.6 [98.9 to 99.9]
  Type 18: n=940 | 91.6 [89.6 to 93.3]

13. Secondary Outcome: Percentage of Original qHPV Vaccine Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 18 Postdose 3 (Month 24)
Description: as for outcome 4
Time Frame: Month 24 (18 Months Post-dose 3)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 595
Percentage of participants
  Type 6: n=446 | 95.1 [92.6 to 96.9]
  Type 11: n=447 | 98.2 [96.5 to 99.2]
  Type 16: n=442 | 98.4 [96.8 to 99.4]
  Type 18: n=447 | 87.5 [84.0 to 90.4]

14. Secondary Outcome: Percentage of Original qHPV Vaccine Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 24 Postdose 3 (Month 30)
Description: as for outcome 4
Time Frame: Month 30 (24 Months Post-dose 3)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 911
Percentage of participants
  Type 6: n=799 | 95.6 [94.0 to 96.9]
  Type 11: n=800 | 97.5 [96.2 to 98.5]
  Type 16: n=795 | 98.6 [97.5 to 99.3]
  Type 18: n=803 | 84.3 [81.6 to 86.8]

15. Secondary Outcome: Percentage of Original qHPV Vaccine Participants Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 31 Postdose 3 (Month 37).
Description: as for outcome 4
Time Frame: Month 37 (31 Months Post-dose 3)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 772
Percentage of participants
  Type 6: n=657 | 94.5 [92.5 to 96.1]
  Type 11: n=657 | 96.0 [94.3 to 97.4]
  Type 16: n=655 | 98.2 [96.8 to 99.0]
  Type 18: n=660 | 81.1 [77.9 to 84.0]

16. Secondary Outcome: Percentage of Participants in the Extension Group Who Are Seropositive for HPV Types 6, 11, 16, and 18 at Month 1 Postdose 3 of qHPV (Month 37)
Description: as for outcome 4
Time Frame: Month 37 (1 Month Post-dose 3 of qHPV)
Population: Per-protocol population: participants without protocol violations who received all 3 qHPV vaccinations, were seronegative to the respective HPV type at Month 30, and had a valid serology result at the specified time for assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 440
Percentage of participants
  Type 6: n=246 | 99.6 [97.8 to 100]
  Type 11: n=246 | 100 [98.5 to 100]
  Type 16: n=246 | 100 [98.5 to 100]
  Type 18: n=255 | 98.8 [96.6 to 99.8]

17. Secondary Outcome: Geometric Mean Titers of Original qHPV Vaccine Cohort for Anti-HPV 6, 11, 16, and 18 at Month 1 Postdose 3 of qHPV Vaccine (Month 7)
Time Frame: Month 7 (1 Month Post-dose 3)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 1082
milliMerck units/mL
  Type 6: n=953 | 929.2 [871.0 to 991.4]
  Type 11: n=954 | 1362.8 [1279.8 to 1451.3]
  Type 16: n=949 | 5512.7 [5109.9 to 5947.2]
  Type 18: n=956 | 1278.9 [1183.2 to 1382.4]

18. Secondary Outcome: Geometric Mean Titers of Original qHPV Vaccine Cohort for Anti-HPV 6, 11, 16, and 18 at Month 12 Postdose 3 of qHPV Vaccine (Month 18)
Time Frame: Month 18 (Month 12 Post-dose 3)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 1106
milliMerck units/mL
  Type 6: n=937 | 219.3 [204.9 to 234.7]
  Type 11: n=938 | 296.9 [276.9 to 318.3]
  Type 16: n=933 | 1314.8 [1220.5 to 1416.5]
  Type 18: n=940 | 203.0 [184.1 to 223.9]

19. Secondary Outcome: Geometric Mean Titers of Original qHPV Vaccine Cohort for Anti-HPV 6, 11, 16, and 18 at Month 18 Postdose 3 of qHPV Vaccine (Month 24)
Time Frame: Month 24 (18 Months Post-dose 3)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Groups:
- qHPV Vaccine in Base Study: Represent participants randomized to the qHPV vaccine group
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 595
milliMerck units/mL
  Type 6: n=446 | 143.5 [129.2 to 159.5]
  Type 11: n=447 | 206.6 [186.9 to 228.3]
  Type 16: n=442 | 932.1 [833.3 to 1042.7]
  Type 18: n=447 | 136.2 [118.5 to 156.6]

20. Secondary Outcome: Geometric Mean Titers of Original qHPV Vaccine Cohort for Anti-HPV 6, 11, 16, and 18 at Month 24 Postdose 3 of qHPV Vaccine (Month 30)
Time Frame: Month 30 (24 Months Post-dose 3)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 911
milliMerck units/mL
  Type 6: n=799 | 146.5 [135.6 to 158.2]
  Type 11: n=800 | 177.0 [163.6 to 191.5]
  Type 16: n=795 | 826.1 [757.8 to 900.5]
  Type 18: n=803 | 114.7 [102.8 to 127.9]

21. Secondary Outcome: Geometric Mean Titers of Original qHPV Vaccine Cohort for Anti-HPV 6, 11, 16, and 18 at Month 31 Postdose 3 of qHPV Vaccine (Month 37)
Time Frame: Month 37 (31 Months Post-dose 3)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 772
milliMerck units/mL
  Type 6: n=657 | 128.6 [118.2 to 139.9]
  Type 11: n=657 | 149.7 [137.0 to 163.6]
  Type 16: n=655 | 680.4 [617.2 to 750.1]
  Type 18: n=660 | 102.4 [90.9 to 115.3]

22. Secondary Outcome: Geometric Mean Titers in the Extension Group for Anti-HPV 6, 11, 16, and 18 at Month 1 Postdose 3 of qHPV Vaccine (Month 37)
Time Frame: Month 37 (1 Month Post-dose 3 of qHPV)
Population: Per-protocol population: participants without protocol violations who received all 3 qHPV vaccinations within appropriate day ranges, were seronegative to the respective HPV type at Month 30, and had a valid serology result at the specified time for assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 440
milliMerck units/mL
  Type 6: n=246 | 768.6 [676.6 to 873.0]
  Type 11: n=246 | 1041.0 [919.8 to 1178.2]
  Type 16: n=246 | 4312.7 [3715.6 to 5005.7]
  Type 18: n=255 | 830.1 [714.0 to 965.1]

23. Secondary Outcome: Combined Incidence of HPV 6/11/16/18-related Persistent Infection and HPV 6/11/16/18-related CIN, AIS, VIN, VaIN, Genital Warts, and Cervical/Vaginal/Vulvar Cancer in Females
Description: The HPV types were determined by polymerase chain reaction (PCR) testing. The combined incidence of HPV 6/11/16/18-related persistent infection and HPV 6/11/16/18-related cervical intraepithelial neoplasia (CIN), adenocarcinoma in situ (AIS), vulvar intraepithelial neoplasia (VIN), vaginal intraepithelial neoplasia (VaIN), genital warts, and cervical/Vaginal/vulvar cancer was assessed in female participants.
Time Frame: Up to Month 126
Population: Per-Protocol Effectiveness population: male participants without protocol violations who received at least 1 dose of qHPV vaccine and at least 1 effectiveness follow-up visit.
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years at risk
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 259 | 96
Cases per 100 person-years at risk | 0.2 [0.1 to 0.7] | 0.2 [0.0 to 1.4]

24. Secondary Outcome: Combined Incidence of HPV 6/11/16/18-related Persistent Infection and HPV 6/11/16/18-related PIN, Genital Warts, and Penile/Perineal/Perianal Cancer in Males
Description: The HPV types were determined by PCR testing. Combined incidence of HPV 6/11/16/18-related persistent infection and HPV 6/11/16/18-related penile/perineal/perianal intraepithelial neoplasia (PIN), genital warts, and penile/perineal/perianal cancer was assessed in male participants.
Time Frame: Up to Month 126
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years at risk
Arm/Group | qHPV Vaccine in Base Study | qHPV Vaccine in Extension Study
Number analyzed (Participants) | 179 | 62
Cases per 100 person-years at risk | 0.6 [0.2 to 1.5] | 0.3 [0.0 to 1.9]

ADVERSE EVENTS:
Time Frame: Day 1 to Month 30 and Month 30 to Month 126
Description: Day 1 to Month 30: All adverse events were collected up to Day 15 after any vaccination. Month 30 to Month 126: Nonserious AEs were not collected. Deaths and related SAEs were collected throughout the study. Non-serious AEs were not solicited during the Extension Study; any reported non-serious AEs were unsolicited and not systematically assessed.
Groups:
- qHPV Vaccine in Base: Vaccine Phase and Follow-up: Participants who were randomized into the qHPV Group, who received three 0.5 mL intramuscular injections of qHPV at Day 1, Month 2, and Month 6, and had safety follow-up. Adverse events are reported for this group from Day 1 to Month 30.
- Placebo in Base: Vaccine Phase and Follow-up: Participants who were randomized into the Placebo Group, who received three 0.5 mL intramuscular injections of placebo vaccine at Day 1, Month 2, and Month 6, and had safety followup.
  Adverse events are reported for this group from Day 1 to Month 30.
- qHPV Vaccine in Base: Extension and Long-term Follow-up: Participants who received qHPV in the Base Study. No study treatment was administered after Month 6 for these participants. Adverse events are reported for this group from Month 30 to Month 126. Non-serious AEs were not solicited.
- qHPV Vaccine in Extension: Extension and Long-term Follow-up: Participants who received placebo in the Base Study and three 0.5 mL intramuscular injections of V501 (qHPV) at Month 30, Month 32, and Month 36 in the Extension Study. Adverse events are reported for this group from Month 30 to Month 126. Non-serious AEs were not solicited.
Arm/Group | qHPV Vaccine in Base: Vaccine Phase and Follow-up | Placebo in Base: Vaccine Phase and Follow-up | qHPV Vaccine in Base: Extension and Long-term Follow-up | qHPV Vaccine in Extension: Extension and Long-term Follow-up
Serious Adverse Events (participants affected / at risk) | 6/1165 | 0/584 | 2/932 | 3/481
Other Adverse Events (participants affected / at risk) | 918/1165 | 344/584 | 0/932 | 3/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine in Base: Vaccine Phase and Follow-up (N=1165) | Placebo in Base: Vaccine Phase and Follow-up (N=584) | qHPV Vaccine in Base: Extension and Long-term Follow-up (N=932) | qHPV Vaccine in Extension: Extension and Long-term Follow-up (N=481)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonic clonic movements (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine in Base: Vaccine Phase and Follow-up (N=1165) | Placebo in Base: Vaccine Phase and Follow-up (N=584) | qHPV Vaccine in Base: Extension and Long-term Follow-up (N=932) | qHPV Vaccine in Extension: Extension and Long-term Follow-up (N=481)
Injection site erythema (General disorders) | 237 (323) | 78 (109) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 853 (1705) | 268 (434) | 0 (0) | 3 (3)
Injection site swelling (General disorders) | 241 (336) | 45 (63) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 100 (114) | 44 (60) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 221 (297) | 111 (163) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 52 (56) | 24 (26) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The difference between the prior and final data is a minor change in the definition of the per-protocol immunogenicity population, which was applied down to the base study. Also, protocol violators were identified and excluded from the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.